CLINICAL TRIAL: NCT02295137
Title: Image Fusion of Pre-procedural CTA With Real-time Fluoroscopy to Guide Proper Renal and Visceral Arteries Catheterization During Advanced Endovascular Aortic Aneurysms Repair: A Feasibility Study
Brief Title: Image Fusion of Preprocedural CTA With Real Time Fluoroscopy to Enhance EVAR Repair
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN
Record Dates: First submitted 2014-10-27; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-10

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pre-procedure image guidance (Experimental)
  Interventions: Procedure: Using pre-procedural CTA to guide advanced EVAR procedure

INTERVENTIONS:
Procedure: Using pre-procedural CTA to guide advanced EVAR procedure

SUMMARY:
Abdominal Aortic Aneurysm (AAA) is a potentially life threatening condition. If the aneurysm ruptures, the mortality can be as high as 80%. Endovascular aneurysms repair (EVAR) is a minimal invasive procedure and has been widely used on treating AAA. Advanced endovascular techniques are used to treat patients with more complex pathology by using custom-made devices and additional stents. In order to accomplish the technical success on advanced EVAR, with the current imaging equipment and technique for EVAR procedures (i.e. live x-ray fluoroscopy and 2-D digital subtraction angiography (DSA)), multiple angiograms on the target arteries (arteriograms) are required. Subsequently patients are exposed to higher dose of contrast and radiation, compared to conventional EVAR. This study is to assess the feasibility of proper visceral and renal arteries catheterization using a 3D model obtained from pre-procedural computed tomographic angiography (CTA), fused with real-time fluoroscopy, without contrast injection or angiographic run-offs thus minimizing the contrast use and patient radiation exposure while achieving procedure success during Advanced EVAR.

ELIGIBILITY:
Inclusion Criteria:

* male or female >= 18 years;
* scheduled for advanced EVAR for abdominal aortic aneurysm.

Exclusion Criteria:

* Pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Procedure success | within 1 day
  Evaluate the technical success of advanced EVAR by using pre-procedural CTA images as guidance

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada